CLINICAL TRIAL: NCT04972513
Title: The Emerging Adulthood Health Project
Brief Title: Impact of E-cigarette Use on the Body
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Megan Roberts, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-20320; NCI-2021-06438 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-29; First posted 2021-07-22 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Oscillometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prevention (survey, breathe tests, biospecimen collection): Participants undergo computer-based spirometry testing, nitric oxide breath testing, airwave oscillometry, and an assessment of endothelial function. Participants will undergo collection of blood. Current e-cigarette users also vape their own e-cigarette device for 30 minutes.
  Interventions: Procedure: Biospecimen Collection; Procedure: Nitric Oxide Breath Test; Procedure: Oscillometry; Procedure: Spirometry; Other: Survey Administration; Procedure: Endothelial function

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
Procedure: Nitric Oxide Breath Test — Undergo nitric oxide breath testing
Procedure: Oscillometry — Undergo airwave oscillometry
Procedure: Spirometry — Undergo spirometry
Other: Survey Administration — Complete survey
Procedure: Endothelial function — Endothelial function will be assessed with the EndoPAT device, which measures changes in pressure from sensors placed on the fingertip

SUMMARY:
This study examines how electronic (e)-cigarette use impacts the body, by studying both users and non-users of e-cigarettes. Early evidence indicates that e-cig users experience adverse health effects. Results of this study may help policy-makers develop standards for different types of tobacco.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Examine the short-term impacts of vaping on pulmonary and respiratory outcomes.

OUTLINE:

Current e-cigarette users will vape their own e-cigarette device ad libitum for 30 minutes; non-users will watch a neutral video for 30 minutes. Before and after the 30 minute vaping [video] session, participants will undergo the following assessments: computer-based spirometry testing, nitric oxide breath testing, airwave oscillometry, and an assessment of endothelial function. Participants will also undergo collection of blood.

ELIGIBILITY:
Inclusion Criteria:

* 75 e-cig users and 75 never-users
* No self-reported diagnosis of lung disease (e.g., coronavirus disease-2019 [COVID-19], pneumonia, cystic fibrosis)
* No history of cardiac event or distress
* Not currently breastfeeding, pregnant, or planning to become pregnant (e-cig users only; will be confirmed via pregnancy test)

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: E-cig (cigarette) users and non-users in Ohio
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Airway inflammation as assessed by exhaled nitric oxide | Procedure will last approximately 3 minutes; the procedure will occur twice during the laboratory session (separated by approximately 60 minutes)
  Exhaled nitric oxide will be measured in parts per billion (ppb)
Airway reactivity as assessed by airwave oscillometry | Procedure will last approximately 3 minutes; the procedure will occur twice during the laboratory session (separated by approximately 60 minutes)
  Airway reactivity will be measured via Tremoflo, which is a well validated measurement of airway reactivity and provides curves of Resistance (R) and Reactance (X)
Respiratory functioning as assessed by a mobile Spirometry device | Procedure will last approximately 3 minutes; the procedure will occur twice during the laboratory session (separated by approximately 60 minutes)
  Spirometry will collect daily data from participants on the relationship between their forced expiratory volume and forced vital capacity (measured as FEV1/FVC).
Endothelial function | Procedure will last approximately 20 minutes; the procedure will occur twice during the laboratory session (separated by approximately 90 minutes)
  Endothelial function will be assessed with the EndoPAT device (unit of measurement = LnRHI).

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Roberts, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu